CLINICAL TRIAL: NCT04330872
Title: An Investigation Into The Impact Of Enteric Coated Of Aspirin In Patients With Newly Diagnosed Ischemic Stroke. Non-randomized Interventional Controlled Clinical Trial.
Brief Title: An Investigation Into The Impact Of Enteric Coated Of Aspirin In Patients With Newly Diagnosed Ischemic Stroke.
Acronym: ECASIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-18-156
Record Dates: First submitted 2020-03-23; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enteric coated Aspirin (Active Comparator): EC aspirin loading dose 300mg followed by 100 mg (2 days).
  The study's total duration is 3 days.
  Interventions: Drug: Enteric Coated Aspirin Tablet
- Plain Aspirin (Placebo Comparator): Dispersible Aspirin loading dose 300mg followed by 75mg tablets (2 days)
  The study's total duration is 3 days.
  Interventions: Drug: Plain Aspirin

INTERVENTIONS:
Drug: Enteric Coated Aspirin Tablet — Study participants will be assigned to receive either EC Aspirin and will be required to continue taking them throughout the study (three days).
  Arms: Enteric coated Aspirin
Drug: Plain Aspirin — Study participants will be assigned to receive either Plain Aspirin and will be required to continue taking them throughout the study (three days).
  Arms: Plain Aspirin

SUMMARY:
Uncertainty remains regarding the impact of enteric-coated (EC) aspirin as it relates to the reduction of CV risk. We hypothesize that EC formulation based on the previous report may blunt aspirin response as evidenced by reduced Thromboxane A2 (TXA 2) levels in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed ischemic stroke who are just about to start aspirin.
2. No prior history of cardiovascular morbidity (including ischemic heart disease, chronic kidney disease, peripheral vascular disease) 3-18- 75 years.

4-Patients with ischemic stroke who underwent reperfusion intervention (catheter-directed thrombolysis and/or thrombectomy) regardless of the time of presentation (i.e within or outside the therapeutic window as the managing stroke deem fit.

Exclusion Criteria:

1. Concomitant antiplatelet therapy (irrespective of the duration of the treatment).
2. Patients on any prostaglandins related medications (non-steroidal anti-inflammatory drugs, misoprostol, and other ant secretory drugs among others).
3. Any salicylate-containing supplements.
4. Patients on the NG tube will be excluded from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Aspirin non-responders. | At "Day 3"
  Aspirin nonresponsiveness is defined as a level of residual serum TXB2 associated with elevated thrombotic risk (<99.0% inhibition or TXB2 >3.1 ng/ml) after 3 daily aspirin doses

SECONDARY OUTCOMES:
Incidence of Gastrointestinal bleeding consequent upon aspirin therapy. | After three daily aspirin doses ( at "Day 3")
  Major and minor GIT bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Derived] Elshafei MN, Imam Y, Alsaud AE, Chandra P, Parray A, Abdelmoneim MS, Obeidat K, Saeid R, Ali M, Ayadathil R, Mohamed MFH, Abdallah IM, Mohammed S, Akhtar N, Danjuma MI. The impact of enteric coating of aspirin on aspirin responsiveness in patients with suspected or newly diagnosed ischemic stroke: prospective cohort study: results from the (ECASIS) study. Eur J Clin Pharmacol. 2022 Nov;78(11):1801-1811. doi: 10.1007/s00228-022-03391-2. Epub 2022 Sep 19. PMID 36121499
- [Derived] Elshafei MN, Imam Y, Mohamed MFH, AlSaud AE, Ahmed MS, Obeidat K, Saeid R, Ali M, Abdallah IM, Parray AS, Danjuma MI. An investigation into the impact of enteric coated of aspirin in patients with newly diagnosed ischemic stroke (ECASIS). Medicine (Baltimore). 2020 May;99(20):e20307. doi: 10.1097/MD.0000000000020307. PMID 32443379